CLINICAL TRIAL: NCT02750137
Title: Ametop - Friend or Foe A Prospective Observational Study of the Incidence of Adverse Reactions With Ametop
Brief Title: Ametop - Friend and Foe A Prospective Study of the Incidence of Adverse Reactions With Ametop
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Angela Tan Yun June, Senior Resident, KK Women's and Children's Hospital
Other Study IDs: 2015/2158
Record Dates: First submitted 2016-04-17; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Adverse Drug Event
Keywords: Tetracaine
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Tetracaine

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tetracaine — Application of Ametop prior to intravenous cannulation
  Other Names: Ametop

SUMMARY:
Ametop was introduced into the formulary as it was deemed more efficacious for intravenous cannulation compared to EMLA. However, the incidences of adverse reactions seemed to be higher compared to other studies. This lead to a prospective observational study to look at the incidence and severity of skin reactions following routine clinical application of Ametop.

DETAILED DESCRIPTION:
Ametop was introduced into the formulary as it was deemed more efficacious for intravenous cannulation compared to EMLA. After several critical incidences of adverse reactions that occurred with its application, a departmental audit was carried out to look at the incidence and severity reactions with its application as well as its outcome on intravenous cannulation. The findings of the departmental audit showed that the incidence of adverse reactions seemed to occur more commonly compared to other studies.

A prospective observational study was carried out to look at the incidence and severity of skin reactions following routine clinical application of Ametop.

This study aims to achieve the following:

1. Investigate the incidence and severity of adverse skin reactions following topical application of Ametop prior to intravenous cannulation
2. Assess the success rate of intravenous cannulation
3. Identify the possible risk factors associated with adverse skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients presenting for surgery from August 2014 to May 2015 who have had Ametop applied prior to intravenous cannulation.

Exclusion Criteria:

* Any patient who did not have Ametop applied or have an intravenous cannula in situ.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Paediatric patients presenting for surgery in KK Women's and Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Incidence of skin reactions with Ametop | October 2014 to May 2015
  looking at the incidence of skin reactions with Ametop - normal, simple erythema, raised erythema, itch, pallor

SECONDARY OUTCOMES:
Risk factors associated with incidence of skin reactions | October 2014 to May 2015
  Looking at possible factors associated with skin reactions - race, duration of application, history of atopy

CONTACTS AND LOCATIONS:
Overall Officials: Angela YJ Tan, MMed, Principal Investigator — KK Women's and Children's Hospital

IPD SHARING:
Plan to Share IPD: No
Data will be protected and not shared.

REFERENCES:
- [Background] Browne J, Awad I, Plant R, McAdoo J, Shorten G. Topical amethocaine (Ametop) is superior to EMLA for intravenous cannulation. Eutectic mixture of local anesthetics. Can J Anaesth. 1999 Nov;46(11):1014-8. doi: 10.1007/BF03013194. PMID 10566919
- [Background] Arrowsmith J, Campbell C. A comparison of local anaesthetics for venepuncture. Arch Dis Child. 2000 Apr;82(4):309-10. doi: 10.1136/adc.82.4.309. PMID 10735838